CLINICAL TRIAL: NCT05285709
Title: Evaluation of Novel Biomarkers in Early Recognition of Acute Kidney Injury After Orthopedic Operations.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Marek Janiak, Principal Investigator, Medical University of Warsaw
Other Study IDs: BIAKOR
Record Dates: First submitted 2022-01-21; First posted 2022-03-18 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Hip Fractures; Acute Kidney Injury
MeSH Terms: conditions — Hip Fractures; Acute Kidney Injury | interventions — Environmental Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine and plasma from centrifuged whole blood after partial analysis of biomarkers
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Biomarker — blood and urine sampling before and after surgery (1-admission to operating ward, 2-leaving operation ward, 1st day postop, 2nd day postop, 5th day postop, or the day patient leaves hospital, whichever is first)
Diagnostic Test: RRI measurement — patients able to cooperate will have renal resistive index measured before and after surgery (admission to operating ward, leaving operating ward)

SUMMARY:
Surgical treatment of hip fracture may be complicated by acute kidney injury. The aim of this study is to investigate whether the investigators can find a better biomarker than creatinine to recognize this problem at an earlier stage.

DETAILED DESCRIPTION:
Extensive orthopedic surgical procedures may have many postoperative complications. One of those, sometimes overlooked, is acute kidney injury. Classically defined by KDIGO criteria as an increase in creatinine concentration, may go by unnoticed due to a late peak in serum concentration of this marker. There is still need for "nephrological troponin" which could easily and with a low margin of doubt identify acute kidney injury.

The investigators have planned a double-center study, in cooperation with the 'Department of Anesthesiology and Intensive Therapy with the Postoperative Subdivision' of the 'Samodzielny Publiczny Szpital Kliniczny im. prof. Adama Grucy CMKP' in Otwock, concentrating on measuring concentration of biomarkers known to indicate acute kidney injury in different situations: Proenkephalin (PENK), Dickkopf-3 (DKK3), circular RNA (circRNA), Liver-type Fatty Acid-binding Protein (L-FABP), Netrin-1, semaphorin 3a, Tissue Inhibitor of Matrix Metalloproteinase-2 (TIMP-2), Insulin-like Growth Factor-binding Protein 7 (IGFBP-7), Retinol-binding Protein-4 (RBP-4) aiming to find a marker, or group of markers that would allow recognition of renal injury at an early stage to help minimize the effect.

Patients aged at least 18 years, with a hip fracture undergoing, either hip alloplasty, or internal fixation, after providing informed consent, will be included. Patients with end stage renal disease will be excluded. Blood and urine samples will be collected at 5 points of time: 1 - after admission to the operating ward, 2 - following surgery, before leaving the operating ward, 3 - on the 1st postoperative day, 4 - on the 2nd postoperative day, 5 - on the 5th postoperative day, or the day the patient leaves hospital, whichever is first. Additionally patients who will be able to cooperate will have a renal resistive index measured using ultrasonography.

Blood collected from patients, not longer than 8 hours after collection will be tested for PENK concentration (Spingotec GmbH, Berlin, Germany), then plasma obtained from this sample after centrifuging will be frozen together with centrifugated samples of urine in -80 degrees Celsius till analysis.

Additionally, if the concentration of PENK is elevated, the same sample will be tested after 8, 12 and 24 hours of staying at room temperature, to define stability of the test from blood sampling till measurement.

30 days after surgery, an attempt to contact the patient or his/her family is going to be made, to check if the patient has developed need for renal replacement therapy or has required hospitalisation due to kidney dysfunction together with a 30 day mortality evaluation.

ELIGIBILITY:
Inclusion Criteria:

* age at least 18 years
* be able to provide informed consent

Exclusion Criteria:

* end stage renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients able to provide informed consent, who do not have diagnosed end stage renal disease undergoing surgical treatment of hip fracture (either joint alloplasty or internal fixation)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Any stage of acute kidney injury as defined by Kidney Diseases Improving Global Outcome | 120 hours
  Concentration of novel biomarkers, its change and change of renal resistive index considering different stages of acute kidney injury

SECONDARY OUTCOMES:
Kidney perfusion evaluated by Renal Resistive Index (RRI) | 48 hours
  Correlation between RRI and concentration of biomarkers
Analysis of proenkephalin concentration | 24 hours
  Change of proenkephalin concentration in the blood sample left at room temperature
Kidney dysfunction and mortality | 30 days
  Evaluation of 30-day need for renal replacement therapy, hospitalization due to kidney failure and/or mortality

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Gruca Orthopaedic and Trauma Teaching Hospital, Otwock, Masovian Voivodeship
  - I Department of Anesthesiology and Intensive Care Warsaw Medical University, Warsaw, Masovian Voivodeship